CLINICAL TRIAL: NCT06439784
Title: Contribution of 99mTc-HDP Whole-body SPECT/CT Imaging by VERITON-CT CZT Camera in Stereotactic Radiotherapy Treatment of Bone Metastases of Prostate Cancer
Brief Title: Contribution of the VERITON-CT Camera in Prostate Bone Radiostereotaxy
Acronym: VERIOS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHB23.06
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Prostatic Cancer
Keywords: whole body SPECT/CT; bone scintigraphy; stereotaxic bone radiation therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- whole body SPEC/CT (Experimental): Patient will endergo whole body SPECT/CT in treatment position
  Interventions: Other: whole body SPECT/CT

INTERVENTIONS:
Other: whole body SPECT/CT — Patient will unergo a whole body SPECT/CT in treatment position

SUMMARY:
Stereotactic radiotherapy enables bone metastases to be treated with highly precise irradiation beams, enabling small targets to be irradiated. Planning requires the use of cross-sectional imaging such as computed tomography (CT) or magnetic resonance imaging (MRI). Bone scintigraphy with Tc99m-labelled biphosphonates (T1/2=6h) is indicated in the extension assessment of prostate cancers. Thanks to the advent of single-photon emission computed tomography (SPECT) based on CZT detectors; whole-body SPECT is now compatible with clinical constraints. We propose to study the value of using whole-body SPECT for planning stereotactic radiotherapy of metastatic prostate cancer. This is a prospective, single-center, non-randomized study involving 30 patients. Patients will benefit from routine examinations (CT scan, MRI) including a bone SPECT/CT in treatment position performed on the VERITON-CT (Spectrum Dynamics, Haifa, Israel). Planning based on whole-body SPECT images will be carried out remotely from the patient's point of care. The examination will be interpreted by the nuclear physician, and planning will be based on the dosimetric CT scanner, as in standard management. Virtual replanning will be carried out at distance from treatment, incorporating SPECT imaging. Treatment plans with and without SPECT will be compared quantitatively and qualitatively. The feasibility of SPECT imaging in the treatment position will be assessed, enabling lesion location imaging and dosimetric scanning to be performed in a single examination. All therapeutic management and clinical follow-up will be carried out as part of routine care.

DETAILED DESCRIPTION:
This is a prospective, single-center, non-randomized study. After a decision in a multidisciplinary consultation meeting, the patient will be offered to join the study. All therapeutic care and clinical follow-up is carried out as part of routine care.

Patients will benefit from routine examinations (CT scan, MRI) including a SPECT/CT scan of the bone in the treatment position. Three hours after injection of 9 MBq/kg of 99mTc-HDP, CT imaging followed by whole-body SPECT/CT will be performed on the VERITON-CT (Spectrum Dynamics, Haifa, Israel). In order to make the images in the treatment position, the molding of the BodyFIX (Elekta) compression system that is used to reposition the patient between sessions will be made on the examination bed of the VERITON. It is a mattress that stiffens due to air vacuums. It will be placed on an external radiotherapy tray as for the dosimetry scanner. If it is not possible to take the images under these conditions, the patient will benefit from an examination in the standard position.

The images will then be interpreted by a nuclear physician who will identify the targets and define the contours from the SPECT/CT data using the segmentation tools available in the Syngo.via visualization software (Siemens Healthineers, Erlangen, Germany). The images and contours will be anonymized in order to allow blind virtual replanning, at least 6 months before the planning. Non-anonymized images alone will be transmitted as a standard examination, but cannot be incorporated into the treatment plan, as is currently the case.

The patient will benefit from a standard dosimetry scanner for treatment planning. The molding of the mattress made during the SPECT/CT scan of the bone will be reused for the dosimetric scanner. The therapeutic procedure will then follow the local protocol and in line with national recommendations. Whole-body SPECT/CT imaging will then be performed at 3 and 6 months on the conventional examination bed. The targets identified during the reference whole-body SPECT/CT will be reused in order to measure the evolution of the SUV quantification.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* Good general health WHO ≤ 1
* Informed and signed consent prior to any specific study procedure.
* Patient affiliated to the social security system
* Bone metastases from prostate cancer
* Indication for bone stereotactic radiotherapy

Exclusion Criteria:

* Presence of active cancer in the previous three years
* Protected adults (under guardianship or curatorship)
* Unable to undergo medical monitoring for geographical, social or psychological reasons
* Unable to decubitus (orthopnea, etc.),
* Hypersensitivity to HDP or to one of the excipients of the radiopharmaceutical.
* History of radiotherapy of the volume to be treated by stereotaxy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Equivalency of the two treatment plans in quantitative terms | 3 years
  Let m1 be the mean of a dosimetric index from whole-body 99mTc-HDP-SPECT/CT imaging and m2 the mean of the same dosimetric index from standard imaging, the null hypothesis will be "H0: m1 ≠ m2" and the alternative hypothesis "H1: m1 = m2". Thus, if we reject the null hypothesis at the risk of 5% then we will highlight the equivalence between m1 and m2. The statistical approach to set up such tests is called TOST and will require the definition of appropriate and relevant equivalence limits.

SECONDARY OUTCOMES:
Equivalency of the two treatment plans in qualitative terms | 3 years
  The consortium of radiation therapists will decide which treatment plan will be most beneficial for the patient. The proportion of patients whose SPECT/CT-based plan was chosen will be an indicator of the qualitative impact that this imaging can have on the treatment plan. This proportion will also be associated with its 95% confidence interval for accuracy.
Feasibility of SPECT/CT imaging in treatment position | day of SPECT/CT
  The number of patients who have been able to benefit from 99mTc-HDP-SPECT/CT imaging in a treatment position usable in dosimetric planning will be the main indicator of feasibility. Depending on the results of the feasibility of this imaging in the treatment position, we can deduce different conclusions: If the feasibility is demonstrated (25/30 patients) and the primary outcome does not show a difference between the two treatment plans, we will conclude that 99mTc-HDP-SPECT/CT imaging in the treatment position can be substituted for the standard simulation CT scanner. If feasibility is not demonstrated and the primary outcome does not show a difference between the two treatment plans, we will conclude that 99mTc-HDP-SPECT /CT imaging in the treatment position does not contribute to dosimetry planning.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Dieudonne, PhD, Study Director — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France